CLINICAL TRIAL: NCT05143593
Title: Species-specific Bacterial Detector for Fast Pathogen Diagnosis of Severe Pneumonia Patients in Intensive Care Uint: a Multicentre, Randomised Controlled Trial
Brief Title: Species-specific Bacterial Detector for Fast Pathogen Diagnosis of Severe Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-260-04
Record Dates: First submitted 2021-10-13; First posted 2021-12-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-05

CONDITIONS: Severe Pneumonia
Keywords: Diagnosis, Pathogen, Pneumonia
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experiment group (Experimental): antibiotics adjustments are made by two experienced doctors immediately when SSBD results are available, and other treatments are equivalent to those in the control group as routinely
  Interventions: Diagnostic Test: results of SSBD are used to guide antibiotics adjustment
- the control group (No Intervention): As routinely, antibiotics adjustmens are guided on the results of conventional culture tests and other clinical parameters by two experienced doctors.

INTERVENTIONS:
Diagnostic Test: results of SSBD are used to guide antibiotics adjustment — secretions from low resipratory will be obtained on day1,day 3 and day7 after enrollment and detected by SSBD at bedside at once. Antibiotics will be adjusted on the results by experienced doctors.
  Arms: the experiment group

SUMMARY:
This study is a multicenter randomized controlled trial. The purpose of this study is to assess the efficacy of Species-specific Bacterial Dector（SSBD）for fast pathogen diagnosis and treatment in patients with severe pneumonia. Several adult ICU units from the hospitals in Jiangsu province participate the study and the hosted unit is the Department of Critical Care Medicine, Affiliated Drum Tower Hospital of Nanjing University Medical College. All patients who met the inclusion criteria are enrolled and randomly assigned either to the experiment group or to the control group, and received empiral antibiotics initially. In the experiment group, secretions from low respiratory tract are detected by SSBD and conventional culture tests simultaneously on day1,day3 and day7 after enrollment, while in the control group conventional culture tests are carried out on the same days. In the experiment group, antibiotics adjustments are made by two experienced doctors immediately when SSBD results are available, and other treatments are equivalent to those in the control group as routinely. Some clinical parameters and outcomes are recorded.

DETAILED DESCRIPTION:
Sepsis is associated with high morbidity and mortality . Adequate antibiotic therapy in time could decrease mortality and reduce the length of stay in ICU for patients with sepsis or septic shock . As reported in the previous study, the mortality rate of patients increased approximately 7.6% for every hour delayed. Therefore, rapid diagnosis of pathogenic microorganisms is crucial for shortening the time of empirical antibiotic therapy and improving the prognosis of patients with sepsis.

Conventional culture test (CCT) is the most commonly used and golden standard identification method of pathogenic microorganisms in most countries. However, it showed two critical limitations: long time-consuming (2-5 days) and low sensitivity (30-50%), which limited the application of this method in the ICU . To overcome this bottleneck, several new tools were developed and showed significant improvement in time consumption and accuracy. Recently, next-generation sequencing (NGS) technology was applied to acquire the entire information of microorganisms and demonstrated great ability in diagnosing rare pathogens. However, the whole process still needs at least 2 days for the full diagnostic report with high cost. On the other hand, NGS provided too much information about microorganisms but only semi-quantification of pathogens, which was hard for most clinical doctors to extract the most important information to determine antibiotic usage. Other new emerging detection techniques designed by BioFire and Curetis are much superior in detection time than these above. However, its original principle was based on nucleotide diversity of conserved genes among species, which could not satisfy the application in the ICU due to potential false-positive results. Therefore, a unique diagnosis tool aimed at faster and more accurate pathogen identification in the ICU was still a great challenge.

Species-specific gene sequences for bacteria are found creatively. Based on these sequences, species-specific Bacterial Dector（SSBD) are designed. By SSBD, accurate and rapid detection of the most common pathogenic bacteria of sepsis could be carried out bedside conveniently in the ICU in 2~3 hours. A multiple-center randomized controlled trial will be conducted in ICU pneumonia patients to evaluate clinical benefits from SSBD.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. Pneumonia with undetermined pathogen and lower respiratory tract specimens can be obtained ;
3. signed informed consent;

Exclusion Criteria:

1. Pregnant women
2. Lactating women
3. Those who specimens of lower respiratory tract cannot be obtained;
4. The main responsibility of infection was not in the lung, but outside the lung;
5. Patients have participated in other clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Improved Acute Physiology and Chronic Health Evaluation score II score | up to 14 days
  Acute Physiology and Chronic Health Evaluation score II score will be assessed and compared on day1, day3, day7, day10 and day14

SECONDARY OUTCOMES:
the therapeutic turnaround time (TTAT) | on day1, day3,day7
  the time from collecting the specimen for the investigation to initiating appropriate treatment on the results available on test1, test2 ,test3 day.
coverage of appropriate antibiotics | on day1, day3,day7
  numbers of patients with appropriate antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, MD, Study Chair — The Affliated Drum Tower Hospital, Medical School of Nanjing University
Locations (6):
- China (6):
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Affliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Nanjin Drum Tower Hospital Group Suqian Hospital, Suqian, Jiangsu
  - Changshu No.1 People's Hospital, Suzhou, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Yixin People's Hospital, Wuxi, Jiangsu

IPD SHARING:
Plan to Share IPD: No